CLINICAL TRIAL: NCT05987150
Title: Variation in Anisotropy of the Spinal Cord Around Apical Region in Patients With Hyperkyphosis: A Pilot Study Using Diffusion Tensor Imaging
Brief Title: Variation in Anisotropy of the Spinal Cord in Patients With Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-398-01
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hyperkyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type A: Type A was defined as a round/oval spinal cord shape with visible cerebrospinal fluid (CSF) between the cord and the apical vertebrae.
  Interventions: Radiation: Variation in anisotropy of the Spinal Cord using diffusion tensor imaging
- Type B: Type B was defined as a round/oval spinal cord shape with no CSF between the apical vertebrae and spinal cord.
  Interventions: Radiation: Variation in anisotropy of the Spinal Cord using diffusion tensor imaging
- Type C: Type C cord was defined as a spinal cord that is fattened/deformed by the vertebral body, with no visible CSF between the apex and the cord.
  Interventions: Radiation: Variation in anisotropy of the Spinal Cord using diffusion tensor imaging

INTERVENTIONS:
Radiation: Variation in anisotropy of the Spinal Cord using diffusion tensor imaging — All examinations were performed on a 3.0-T MRI machine with a 12-channel spine special coil (Ingenia CX, Philips Healthcare, Best, the Netherlands). The multi-sequence MRI protocol included conventional T1-weighted (sag & tra), T2-weighted (sag & tra), and DTI sequence.

SUMMARY:
Spinal cord compression is commonly seen in patients with severe kyphosis. However, conventional morphologic magnetic resonance imaging (MRI) was unable to detect the damage in microstructural integrity of the spinal cord around the apical vertebrae in these patients. The aim of the study was to evaluate the neuronal metrics/microstructure of the spinal cord around apical region in patients with hyperkyphosis using diffusion tensor imaging (DTI).

DETAILED DESCRIPTION:
Spinal cord compression is commonly seen in patients with severe kyphosis. However, conventional morphologic magnetic resonance imaging (MRI) was unable to detect the damage in microstructural integrity of the spinal cord around the apical vertebrae in these patients. The aim of the study was to evaluate the neuronal metrics/microstructure of the spinal cord around apical region in patients with hyperkyphosis using diffusion tensor imaging (DTI).

Twenty-four patients with hyperkyphosis aged 46.1±22.8 years who underwent 3.0T MRI examination with DTI sequence were prospectively enrolled from July 2022 to January 2023. Patients were divided into three groups according to spinal cord/cerebrospinal fluid architecture (CSF) on sagittal-T2 MRI of the thoracic apex: Type A-circular cord with visible CSF, Type B-circular cord but no visible CSF at apical dorsal, and Type C-spinal cord deformed without intervening CSF. The Fractional Anisotropy (FA) values acquired from DTI were compared among different groups. Correlations between DTI parameters and global kyphosis (GK)/sagittal deformity angular ratio (SDAR) were evaluated using Pearson correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hyperkyphosis;
* the apex located at the thoracal region (T1-T12);
* full DTI data;
* records of detailed and systematic neurological physical examination.

Exclusion Criteria:

* any case with active infection, tumor, or trauma;
* any cases of comorbidity of neurofibromatosis type I;
* any cases combined with spinal syringomyelia, split cord malformations or diastematomyelia, tethered cord syndrome;
* previous spinal surgery.

Ages: 11 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 24 patients with hyperkyphosis aged 46.1±22.8 years who underwent 3.0T magnetic resonance imaging (MRI) examination with DTI sequence were prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy (FA) values | preoperative
  Raw DTI data were postprocessed on FuncTool (GE) software. After an initial correction of geometric distortions, the color-coded FA maps were generated.

SECONDARY OUTCOMES:
Global kyphosis (GK) in degrees | preoperative
  Measured on anteroposterior and lateral radiographs and defined as the angle from upper to lower most tilted end vertebrae.
Sagittal deformity angular ratio (SDAR) | preoperative
  Divided GK by the number of levels spanning the curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No